CLINICAL TRIAL: NCT02417285
Title: A Phase 1b Open-label Study to Evaluate the Safety and Efficacy of CC-122 in Combination With Obinutuzumab (GA101) in Subjects With Relapsed/Refractory Diffuse Large B-Cell Lymphoma and Indolent Non-Hodgkin's Lymphoma
Brief Title: A Phase 1b Open-label Study to Evaluate the Safety and Efficacy of CC-122 With Obinutuzumab (GA101) in Relapsed/Refractory DLBCL and iNHL.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-122-NHL-001
Record Dates: First submitted 2015-04-10; First posted 2015-04-15 (Estimated); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin
Keywords: Non-Hodgkin's Lymphoma; Diffused Large B-Cell Lymphoma; Phase 1B; Open-Label; Safety and Efficacy; CC-122; Obinutuzumab; GA101; Relapsed; Refractory
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Recurrence | interventions — obinutuzumab; 3-(5-amino-2-methyl-4-oxoquinazolin-3(4H)-yl)piperidine-2,6-dione

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CC-122 in combination with Obinutuzumab (Experimental): CC-122 will be administered orally QD starting on Day 1 for 5 consecutive days followed by 2 days off study drug every 7 days (5/7-day schedule) in each 28-day cycle in combination with Obinutuzumab administered as an intravenous (IV) infusion at a dose of 1000 mg on Days 2, 8, and 15 of Cycle 1 and on Day 1 of Cycles 2 through 8.
  Interventions: Drug: Obinutuzumab; Drug: CC-122

INTERVENTIONS:
Drug: Obinutuzumab — 1000 mg administered IV on Days 2, 8, and 15 of Cycle 1 and on Day 1 of Cycles 2 though 8.
  Other Names: GA-101
Drug: CC-122 — CC-122 1mg, 2mg, 3mg, 4mg or 5mg administered orally once daily on a 5/7-day schedule in each 28-day cycle. In addition, subjects will be enrolled on the CC-122 formulated capsule (F6) and evaluated for safety and tolerability in combination with GA101 (Obinituzumab) in a separate cohort. The CC-122 dose will be escalated until the MTD is established on the CC-122 formulated capsule (F6) in combination with GA101 (Obinituzumab).

SUMMARY:
CC-122-NHL-001 study is a multicenter, open-label, phase Ib study with dose escalation and expansion parts. It evaluates the safety, tolerability and clinical pharmacokinetics of CC-122 in combination with obinutuzumab (GA101). The study is also assessing the preliminary efficacy of the combination as well as pharmacodynamic and tumor biomarkers as exploratory objectives. In the dose escalation part, the safety and tolerability of increasing doses of CC-122 administered with a fixed dose of obinutuzumab will be administered to identify the maximum tolerated dose. In the dose expansion part, more patients will be enrolled at a CC-122 dose selected from the escalation part of the study in combination with fixed dose obinutuzumab to further study safety and efficacy.

DETAILED DESCRIPTION:
The one or two cohorts during the dose expansion phase (Part B) will enroll subjects with relapsed or refractory follicular lymphoma (FL) who were either refractory to or relapsed after treatment with a lenalidomide-containing regimen (FL-1 cohort) or never been exposed to lenalidomide (FL-2 cohort). The FL-1 and FL-2 cohorts will enroll up to 20 and/or up to 30 subjects, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures are conducted.
2. ≥ 18 years of age or older at the time of signing the informed consent document.

   Entry Criteria Specific for Dose-Escalation Phase (Part A)
3. Subjects with CD20 positive, histologically or cytologically-confirmed, diffuse large B-cell lymphoma (DLBCL)(including transformed low grade lymphoma) who have relapsed or refractory disease following at least two prior standard treatment regimens (eg, R-CHOP or similar first-lineregimen and at least one second-line salvage regimen) and/or autologous stem cell transplant (ASCT) in chemotherapy-sensitive patients, with the following ASCT

   EXCEPTIONS:
   * Subjects in the pre-ASCT setting with poor prognosis, defined as primary refractory disease, that have relapsed within 12 months following first-line treatment; "double-hit" lymphomas with Bcl-2/Myc gene rearrangements or, overexpression or high IPI score (2,3) at relapse.
   * Subjects refusing ASCT or for whom ASCT is not appropriate based on the Investigator's judgment.

   Entry Criteria Specific for Dose-Expansion Phase (Part B)
4. Subjects with CD20 positive, histologically confirmed (by WHO 2008 classification [Jaffe, 2009]), FL (Grade 1, 2, or 3a) who have relapsed or refractory disease following at least one prior standard systemic treatment regimen including systemic chemo-, immune-, or chemoimmunotherapy.

   Systemic therapy includes treatments such as rituximab monotherapy, chemotherapy given with or without rituximab, radio-immunoconjugates such as 90Y-ibritumomab tiuxetan and 1311-tositumomab. Systemic therapy does not include, for example, H. pylori eradication or antibiotic treatment.

   Lenalidomide naïve
   1. Relapsed or refractory follicular lymphoma (Grade 1, 2, or 3a) following at least one prior standard systemic treatment regimen including systemic chemo-, immune-, or chemoimmunotherapy with no prior exposure to lenalidomide (FL-1 cohort)

      Lenalidomide exposed
   2. Relapsed or refractory follicular lymphoma (Grade 1, 2, or 3a) previously treated with at least two cycles of lenalidomide-containing regimen (FL-2 cohort), either as a single agent or in combination, and experienced outcomes to the lenalidomide treatment as follows:

   Early relapse after lenalidomide treatment: Subjects with relapse within one year of last dose of lenalidomide (or a lenalidomide-containing regimen) following initial response of Complete Response (CR) to lenalidomide (or a lenalidomide-containing regimen) Early progression after lenalidomide treatment: Subjects with Progressive Disease (PD) within one year of last dose of lenalidomide (or lenalidomide-containing regimen) following initial response of partial response (PR) to lenalidomide (or a lenalidomide-containing regimen) Disease refractory to lenalidomide: Subjects with best response of stable disease (SD) or PD while on lenalidomide (or lenalidomide-containing regimen) without any documented response of PR or better during treatment with lenalidomide (or a lenalidomide-containing regimen) Lenalidomide or lenalidomide - containing regimen does not need to be the immediate prior regimen received by the subject to be eligible for entry.

   Entry Criteria that apply to both Part A and Part B
5. Subjects with CD20 positive, histologically confirmed (by WHO 2008 classification [Jaffe, 2009]), FL (Grade 1, 2, or 3a) who have relapsed or refractory disease following at least one prior standard systemic treatment regimen including systemic chemo-, immune-, or chemoimmunotherapy.

   Systemic therapy includes treatments such as rituximab monotherapy, chemotherapy given with or without rituximab, radio-immunoconjugates such as 90Y-ibritumomab tiuxetan and 1311-tositumomab. Systemic therapy does not include, for example, H. pylori eradication or antibiotic treatment.

   Lenalidomide naïve
   1. Relapsed or refractory follicular lymphoma (Grade 1, 2, or 3a) following at least one prior standard systemic treatment regimen including systemic chemo-, immune-, or chemoimmunotherapy with no prior exposure to lenalidomide (FL 2 cohort). In addition, subjects must have received one prior line of salvage therapy, unless ineligible for autologous transplant.

      Lenalidomide exposed
   2. Relapsed or refractory follicular lymphoma (Grade 1, 2, or 3a) previously treated with at least two cycles of lenalidomide-containing regimen (FL-1 cohort), either as a single agent or in combination, and experienced outcomes to the lenalidomide treatment as follows:

   Early relapse after lenalidomide treatment: Subjects with relapse within one year of last dose of lenalidomide (or a lenalidomide-containing regimen) following initial response of Complete Response (CR) to lenalidomide (or a lenalidomide-containing regimen) Early progression after lenalidomide treatment: Subjects with Progressive Disease (PD) within one year of last dose of lenalidomide (or lenalidomide-containing regimen) following initial response of partial response (PR) to lenalidomide (or a lenalidomide-containing regimen) Disease refractory to lenalidomide: Subjects with best response of stable disease (SD) or PD while on lenalidomide (or lenalidomide-containing regimen) without any documented response of PR or better during treatment with lenalidomide (or a lenalidomide-containing regimen) Lenalidomide or lenalidomide - containing regimen does not need to be the immediate prior regimen received by the subject to be eligible for entry.

   Entry Criteria that apply to both Part A and Part B
6. Bi-dimensionally measurable disease on cross sectional imaging by Computed Tomagraphy (CT) or Magnetic resonance imaging (MRI) with at least one lesion > 1.5 cm in the transverse diameter, as defined by the International Working Group (IWG) NHL criteria

   Measurable disease cannot be previously irradiated.
7. ECOG PS (Eastern Cooperative Oncology Group Scale of Performance Status) of 0 to 1.
8. Subjects must have the following laboratory values at screening:

   * Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L without growth factor support for 7 days (14 days if subject received pegfilgrastim).
   * Hemoglobin (Hgb) ≥ 8 g/dL.
   * Platelets (plt) ≥ 50 x 109/L without transfusion for 7 days.
   * Potassium within normal limits or corrected with supplements.
   * Aspartate aminotransferase/Serum glutamic-oxaloacetic transaminase (AST/SGOT) and Alanine aminotransferase / Serum glutamic pyruvic transaminase (ALT/SGPT) ≤ 2.5 x Upper Limit of Normal (ULN) or ≤ 5.0 x ULN if liver tumor is present.
   * Serum bilirubin ≤1.5 x ULN except in cases of Gilberts Syndrome, then ≤ 2.0 x ULN
   * Estimated serum creatinine clearance of ≥ 60 mL/min using the Cockcroft-Gault equation.
9. Per the Pregnancy Prevention Risk Management Plan (PPRMP)

   1. Females of childbearing potential (FCBP) must undergo pregnancy testing based on the frequency outlined in PPRMP and pregnancy results must be negative.
   2. Unless practicing complete abstinence from heterosexual intercourse, sexually active FCBP must agree to use adequate contraceptive methods as specified in PPRMP.

      Complete abstinence is only acceptable in cases where this is the preferred and usual lifestyle of the subject.

      Periodic abstinence (calendar ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable.
   3. Males (including those who have had a vasectomy) must use barrier contraception (condoms) when engaging in sexual activity with FCBP as specified in PPRMP.
   4. Males must agree not to donate semen or sperm for the duration specified in PPRMP.
   5. All subjects must:

      Understand that the study drugs could have a potential teratogenic risk. Agree to abstain from donating blood while taking study drugs and following discontinuation of investigational product.

      Agree not to share study drugs with another person.
   6. Other than the subject, FCBP and males able to father a child should not handle the study drugs or touch the capsules, unless gloves are worn.
   7. Be counseled about pregnancy precautions and risks of fetal exposure (refer to PPRMP, Appendix B)
10. Able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
2. Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
3. Any condition that confounds the ability to interpret data from the study.
4. Symptomatic central nervous system involvement.
5. Any history of progressive multifocal leukoencephalopathy (PML).
6. Known symptomatic acute or chronic pancreatitis.
7. Persistent diarrhea or malabsorption ≥ NCI CTCAE Grade 2, despite medical management.
8. Peripheral neuropathy ≥ NCI CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events) Grade 2
9. Impaired cardiac function or clinically significant cardiac diseases, including any of the following:

   * LVEF (left ventricular ejection fraction) < 45% as determined by MUGA (multi-gated acquisition scan) or ECHO (echocardiogram).
   * Complete left bundle branch or bifascicular block.
   * Congenital long QT syndrome.
   * Persistent or clinically meaningful ventricular arrhythmias.
   * QTcF > 460 msec on Screening ECG (electrocardiogram) (mean of triplicate recordings as assessed by central read).
   * Unstable angina pectoris or myocardial infarction ≤ 6 months prior to starting study drugs.
   * Troponin T value > 0.4 ng/mL or BNP > 300 pg/mL
   * Subjects with baseline troponin T > ULN or BNP > 100 pg/mL are eligible but must have a cardiologist evaluation prior to enrollment in the trial for baseline assessment and optimization of cardioprotective therapy.
10. Prior ASCT (autologous stem cell transplant) ≤ 3 months before first dose.
11. Prior allogeneic stem cell transplant with either standard or reduced intensity conditioning.
12. Prior systemic cancer-directed treatments or investigational modalities ≤ 5 half lives or 1 month prior to starting study drugs, whichever is shorter
13. Prior radiotherapy within 1 month prior to starting study drugs.
14. A major surgery ≤ 2 weeks prior to starting study drugs. Subjects must have recovered from any effects of recent surgery or therapy that might confound the safety evaluation of study drug.
15. Prior treatment with CC-122
16. History of severe allergic or anaphylactic reactions to humanized monoclonal antibodies.

    a. Allergic to any excipients in obinutuzumab.
17. Known human immunodeficiency virus (HIV) infection.
18. Known chronic active hepatitis B or C virus (HBV, HCV) infection.

    1. Subjects who are seropositive due to HBV vaccination are eligible.
    2. Subjects who have no active viral infection and are under adequate prophylactics against HBV re-activation are eligible.
19. Need for current chronic systemic corticosteroid therapy (≥ 10 mg of prednisone per day or an equivalent dose of other anti-inflammatory corticosteroids).

    a. Stable use of inhaled corticosteroids is allowed.
20. Treatment-related myelodysplastic syndrome.
21. Prior history of secondary malignancies (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast) unless the subject has been free of the disease for ≥ 1 year prior to starting study drugs.
22. Prior immunization with live virus vaccines (within 3 months prior to starting study drug) or anticipated immunization with live virus vaccines during the duration of the study.
23. Pregnant or nursing females.
24. Unwilling or unable to comply with the protocol, in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-05-22 (Actual); Primary Completion 2019-05-27 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | Approximately 6 years
  Number of participants with adverse events

SECONDARY OUTCOMES:
Tumor Response | Approximately 6 years
  Percentage of subjects with complete response (CR) or partial response (PR) Tumor response will be determined by the Investigator, based on modification of the modified International Working Group (IWG) Response Criteria for Malignant Lymphoma (Cheson,2007) criteria, and summarized using frequency tabulation by dose cohort and tumor type.
Response Duration | Approximately 6 years
  Duration from the time when criteria for response (CR or PR) are met to disease relapse/progression using modified IWG evaluation criteria.
Progression-free Survival (PFS) | Approximately 6 years
  Number of participants who survive without disease progression/relapse (using modified IWG evaluation criteria) or death as a result of any cause and time from the first dose date to disease progression/relapse or death, whichever occurs first
Pharmacokinetics - Cmax | up to 8 months
  Maximum Observed Concentration in plasma
Pharmacokinetics AUC | Up to 8 months
  Area under the Concentration-time Curve
Pharmacokinetics Tmax | Up to 8 months
  Time to Maximum Concentration
Pharmacokinetics T1/2 | Up to 8 months
  Terminal half-life (t1/2)
Pharmacokinetics - CL/F | Up to 8 months
  Apparent total body clearance
Pharmacokinetics - Vz/f | Up to 8 months
  Apparent volume of distribution

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (8):
- France (4):
  - Local Institution - 105, Borddeaux Cedex
  - Local Institution - 102, Marseille
  - Local Institution - 103, Pierre-Bénite
  - Local Institution - 101, Villejuif
- Italy (2):
  - Local Institution - 301, Bologna
  - Local Institution - 302, Torino
- Netherlands (2):
  - Local Institution - 201, Amsterdam
  - Local Institution - 202, Rotterdam

REFERENCES:
- [Derived] Michot JM, Bouabdallah R, Vitolo U, Doorduijn JK, Salles G, Chiappella A, Zinzani PL, Bijou F, Kersten MJ, Sarmiento R, Mosulen S, Mendez C, Uttamsingh S, Pourdehnad M, Hege K, Chen T, Klein C, Hagner PR, Nikolova Z, Ribrag V. Avadomide plus obinutuzumab in patients with relapsed or refractory B-cell non-Hodgkin lymphoma (CC-122-NHL-001): a multicentre, dose escalation and expansion phase 1 study. Lancet Haematol. 2020 Sep;7(9):e649-e659. doi: 10.1016/S2352-3026(20)30208-8. Epub 2020 Aug 3. PMID 32758434
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com